CLINICAL TRIAL: NCT02622867
Title: Nutritional Intervention Clinical Trial to Evaluate the Lactobacillus Plantarum 3547 Probiotic Effects Over Different Inflammation and Immune System Markers in a Group of Healthy Middle-aged People
Brief Title: Lactobacillus Plantarum 3547 Effects Over Inflammatory and Immunologic Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Creaciones Aromáticas Industriales S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lactobacillus plantarum 3547
Record Dates: First submitted 2015-11-18; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: VOLUNTEERS
Keywords: Lactobacillus plantarum; Maltodextrin; Probiotics; Randomized Controlled Trial
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus plantarum 3547 (Experimental): 1 capsule/daily during 12 weeks with Lactobacillus plantarum 3547 (10x109 cfu/d). The capsule contains 77 mg probiotic Lp3547 and 390 mg maltodextrin
  Interventions: Other: Lactobacillus plantarum 3547
- Maltodextrin (Placebo Comparator): 1 daily capsule of maltodextrin (425 mg) during 12 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Other: Lactobacillus plantarum 3547 — During one period of parallel study (12 weeks) volunteers consumed 1 capsule/daily with Lactobacillus plantarum 3547 immediately after finishing their meal.
  Arms: Lactobacillus plantarum 3547
Dietary Supplement: Maltodextrin — During one period of parallel study (12 weeks), volunteers will consume 1 daily capsule of maltodextrin immediately after finishing their meal.
  Arms: Maltodextrin

SUMMARY:
The purpose of this study is to evaluate the effects of the probiotic Lactobacillus plantarum 3547 over different inflammation and immune system markers on a healthy middle-aged group.

DETAILED DESCRIPTION:
In this randomized double blind controlled trial, a group of healthy middle-aged people (45 to 65 years old) had a nutritional intervention to evaluate the Lactobacillus plantarum 3547 probiotic effects over different inflammation and immune system markers, the experimental group took the experimental supplement (Lactobacillus plantarum 3547) during one period of parallel study (12 weeks), the volunteers consumed 1 capsule/daily with Lactobacillus plantarum 3547 (10x109 cfu/d) immediately after finishing their meal, the capsule contains: 77 mg probiotic Lp3547 and 390 mg maltodextrins. The control group took the control supplement (Maltodextrin) during one period of parallel study (12 weeks), volunteers consumed 1 daily capsule of maltodextrin without Lactobacillus plantarum 3547 (Placebo) immediately after finishing their meal. (The capsule contains 425 mg of maltodextrin)

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 45 to 65 years old;
* Body Mass Index (BMI) ≥ 18,5 and < 40 kg/m2
* Signed informed consent.
* Adequate cultural level and understanding for the clinical trial.
* Free of infections at baseline

Exclusion Criteria:

* Individuals with severe diseases (hepatic, kidney, cancer…);
* Individuals with diagnosed metabolic syndrome, diabetes and/or hyperthyroidism;
* Individuals with chronic intestinal pathologies (Gastritis, Colitis, Irritable Bowel Syndrome, Pseudomembranous Colitis, Crohn's disease…);
* Individuals with dementia, mental disease or low cognitive function;
* Individuals with autoimmune diseases and/or under treatment with corticosteroids and/or immunosuppressants;
* Individuals with major surgeries during the last month or gastrointestinal surgery in the last 3 months;
* Individuals treated with oral antibiotics during two weeks prior to the beginning of the study;
* Individuals undergoing dietary restriction and/or pharmacological treatment for the decrease of body weight 2 months prior to the beginning of the study;
* Individuals who intend to quit smoking during the next 20 weeks;
* Women that consume oral contraceptive;
* Pregnant women or breastfeeding;
* Individuals with intensive physical activity (> 2 hours, more than 3 times per week);
* Individuals that consume antioxidant supplement, drugs, ω-3 supplements, vitamins, minerals, prebiotics or/and probiotics during the 2 weeks prior to the beginning of the study and that will not eliminate their consumption during the study;
* Individuals with regular consumption (> 3 servings per week) of fermented foods (yogurt, actimel, kefir, blue cheese…) and/or use of other prebiotics and not to accept suppress their consumption during the study;
* Individuals with increased alcohol consumption >30g/day (equivalent to 300 ml of wine, about 3 beers or a cup (75 ml) of whiskey , brandy , anise, etc);
* Individuals with regular use of laxatives (> 2 a week) and (Laxbene, Miralax, Dulco - Lax, etc.) and does not accept suppress its consumption during the study period.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline interleukin 6 (IL-6) | 0 and 12 weeks
Change from baseline interleukin 1β (IL1β) | 0 and 12 weeks
Change from baseline interleukin 10 (IL10) | 0 and 12 weeks
Change from baseline cytokine Tumor necrosis factor (TNFα) | 0 and 12 weeks
Change from baseline Mcp1 (Monocyte Chemoattractant Protein-1) | 0 and 12 weeks
Transforming growth factor beta 1 (TGF-β1) | 0 and 12 weeks
Change from baseline Interferon gamma (INF-γ) | 0 and 12 weeks

SECONDARY OUTCOMES:
Change from baseline cluster of differentiation 4 "CD4+T cells" | 0 and 12 weeks
Change from baseline T lymphocytes | 0 and 12 weeks
Change from baseline cluster of differentiation 8 "CD8+ T cells" | 0 and 12 weeks
Change from baseline natural killer cells | 0 and 12 weeks
Change from baseline B lymphocytes | 0 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, MD, PhD, Principal Investigator — La Paz University Hospital
Locations (1):
- La Paz University Hospital, Madrid, Madrid, Spain

REFERENCES:
- See also: La Paz University Hospital Research Institute — http://www.idipaz.es/